CLINICAL TRIAL: NCT02651974
Title: Evidence Based Colorectal Cancer Screening for the Uninsured - Sub-study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 082012-086 Sub-study
Record Dates: First submitted 2015-11-02; First posted 2016-01-11 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer
Keywords: neoplasm; colorectal; cancer; uninsured; FIT; fecal immunochemical test
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control condition (Active Comparator): A control invitation letter similar to the previous standard (non-incentive) invitation with slight wording and grammatical improvements will be mailed to patients randomly assigned to this group.
  Interventions: Behavioral: Cost condition; Behavioral: Cost/Future condition
- Cost condition (Active Comparator): A control invitation letter with the addition of one line informing participants of the average value of the KIT procedure will be mailed to patients randomly assigned to this group.
  Interventions: Behavioral: Control condition; Behavioral: Cost/Future condition
- Cost/Future condition (Active Comparator): An invitation letter with the average value of the KIT procedure and a sentence assuring participants that should a follow-up test be requested, it will also be provided free of charge will be mailed to patients randomly assigned to this group.
  Interventions: Behavioral: Control condition; Behavioral: Cost condition

INTERVENTIONS:
Behavioral: Control condition — Patients will be mailed a control invitation letter to complete a home fecal immunochemical test (FIT) for colorectal cancer screening.
  Arms: Cost condition; Cost/Future condition
Behavioral: Cost condition — Patients will be mailed a cost condition invitation letter to complete a home fecal immunochemical test (FIT) for colorectal cancer screening.
  Arms: Control condition; Cost/Future condition
Behavioral: Cost/Future condition — Patients will be mailed a cost/future condition invitation letter to complete a home fecal immunochemical test (FIT) for colorectal cancer screening.
  Arms: Control condition; Cost condition

SUMMARY:
This is a sub-study nested within a previously initiated clinical study (# NCT01946282) focusing on individuals not previously randomized at baseline to the original interventions. The purpose of the sub-study is to evaluate, via a randomized controlled trial design, 3 strategies for promoting screening completion among individuals not up to date with colorectal cancer screening, but assigned to receive screening outreach.

DETAILED DESCRIPTION:
In the previously initiated, ongoing clinical study (# NCT01946282) investigators are testing a systematic colon cancer screening outreach strategy for increasing screening completion among uninsured patients, not up-to-date with screening. This is a Sub-study to #NCT01946282 (IRB # 082012-086).

Sub-study description:

The goal of the sub-study is to identify strategies that may further increase rates of 1) initial participation in colorectal cancer screening, and 2) follow up of abnormal colorectal cancer screening tests with colonoscopy.

At the time of the sub-study, all patients randomly assigned to receive gift card incentives have been enrolled. At this time only standard, non-incentive invitations continue to be mailed to eligible patients.

The sub-study involves 2 parts:

Part 1: Participants scheduled to receive mailed fecal immunochemical test (FIT) outreach for the first time late in the 2nd year of the study will be randomly assigned to receive one of three invitation letters, which vary slightly from one another.

For the sub-study, the standard invitation letter will be replaced with one of the three sub-study letters. All new participants will receive one of the 3 letters during 2 predetermined rounds of invitations (involving n=2,124 individuals). There will be 3 conditions for the sub-study letters and individuals will be randomly assigned 1:1:1 to each condition. The 3 conditions are as follows:

i) Condition 1 - control letter will be similar to the previous study letters with some slight wording and grammatical improvements, ii) Condition 2 - cost letter will be the control letter plus the addition of one sentence informing recipients of the average value of the FIT procedure and; iii) Condition 3 - cost/future letter will include the average value of FIT and a sentence assuring patients that should a follow-up test be requested, it will be provided free of charge.

Rationale and plan for sub-study Part 1: Over nearly 2 years of the program the investigators have tested a systematic outreach strategy for increasing screening completion among uninsured patients, not up to date with screening. Through these carefully evaluated interventions, the investigators have shown that an outreach invitation strategy, particularly when it includes FIT invitations, markedly increases screening completion among the uninsured. Thirty-six percent of individuals invited to complete FIT return the test. The investigators believe this rate may be improved by making changes to the invitation letters. The sub-study hypothesis is that providing information in the letter about the value of the kit and attenuating concern about future cost will further increase FIT and follow-up response rates.

Part 2: In part 2 of the sub-study, participants will receive their FIT results in either a white envelope (normal results, no immediate follow-up necessary) or a red envelope (abnormal result, need to follow-up with physician). The only change to this portion of the study is the color of the envelope patients receive.

Rationale and plan for Part 2: With the current program, the rate of follow-up diagnostic colonoscopy after abnormal FIT is 58%. Since individuals with abnormal FIT have an increased chance of having colorectal cancer, identifying alternate strategies to improve compliance with diagnostic colonoscopy is desirable. Accordingly the sub-study will employ a simple alerting tactic through the color of the envelope (red for abnormal and white for normal). The investigators hypothesize that more patients will follow-up after receiving a positive FIT result as a result of the messaging importance of abnormal tests with a red envelope. Because the sub-study will be employed in 2 predetermined rounds of invitations, investigators will have the opportunity to conduct a pre-post analysis of the follow-up rates to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Uninsured
* Participants in John Peter (JPS) Health System medical assistance program for the uninsured.
* One or more visits to a JPS primary care clinic within a year.
* Not up-to-date with colorectal cancer screening

Exclusion Criteria:

* Patients with a history of colorectal cancer or colon resection
* No address and/or phone number on file with JPS
* Incarcerated

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8565 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Percentage of individuals who complete FIT screening measured by return FIT kit | Within 3 months of invitation
  The primary outcome will be analyzed using an intention to treat approach. An "a priori" estimated sample size is 2,124; assigned 1:1:1 via simple randomization, stratified by round of invitation to each of the three intervention groups. Sample size was constrained by the number of individuals eligible for screening outreach; all eligible individuals during study period will be included in one of the intervention groups. Assuming a standard intervention group FIT completion rate of 36%, and two-sided alpha=0.125 for each comparison, an estimated 80% power to detect a >8% difference between Condition 1 (standard mailed invitation, n=708) and Condition 2 (n=708), as well as 80% power to detect a >8% difference between Condition 1 (n=708) and Condition 3 (n=708).

SECONDARY OUTCOMES:
Percentage of individuals who receive a positive (abnormal) FIT result that then call to receive additional information about potential follow-up test. | Within 6 months of mailed FIT results letter
Percentage of individuals who schedule a pre-operative clinic visit (if recommended). | Within 6 months of mailed FIT results letter
Percentage of individuals who complete a colonoscopy (if recommended). | Within 6 months of mailed FIT results letter
Pre-post analysis of current results reporting strategy (which will utilize a white envelope for normal results, and a red envelope for abnormal results) to prior generic envelope for FIT result reporting for both normal and abnormal results. | Within 6 months of mailed FIT results letter
  This will be measured by proportion of individuals with abnormal FIT completing diagnostic colonoscopy pre and post the envelope intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Keith E Argenbright, MD, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: Undecided